CLINICAL TRIAL: NCT03910725
Title: Electrophysiological Remodelling Secondary to Metabolic, Inflammatory and Cardiomyopathic Processes
Brief Title: Electrophysiological Phenotyping Of Patients at Risk of Ventricular Arrhythmia and Sudden Cardiac Death
Acronym: EPORVA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 19HH4965
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Arrhythmia; Sudden Cardiac Death; Cardiomyopathy, Dilated; Obesity; Inflammation
Keywords: Arrhythmia; Cardiomyopathy, Dilated; Electrocardiographic imaging
MeSH Terms: conditions — Arrhythmias, Cardiac; Death, Sudden, Cardiac; Cardiomyopathy, Dilated; Obesity; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obesity: Patients with BMI >40 awaiting stapled bariatric surgery, without a history of or concomitant ischaemic or structural heart disease, arrhythmia or receiving anti-arrhythmic medication, will be recruited prospectively from the bariatric surgery preoperative assessment clinics.
  Interventions: Other: Electrocardiographic imaging
- Rheumatoid arthritis: Patients with RA without diagnosed or known ischaemic or structural heart disease, arrhythmia or receiving anti-arrhythmic medication will be recruited prospectively from rheumatology clinics, prior to initiation of biologic or diseased modifying anti-rheumatic drugs.
  Interventions: Other: Electrocardiographic imaging
- Dilated cardiomyopathy: TTNtv-positive and -negative DCM patients from the Royal Brompton Hospital biobank have provided informed consent to be contacted for research
  Interventions: Other: Electrocardiographic imaging

INTERVENTIONS:
Other: Electrocardiographic imaging — ECGi is a non-invasive body surface mapping technique that collects electrocardiographic data using 252 leads, and combines it with subject specific anatomic data acquired from cross sectional imaging to recreate epicardial electrograms.

SUMMARY:
Obesity, rheumatoid arthritis (RA) and gene-specific dilated cardiomyopathy (DCM) are common medical conditions. Small-scale studies have shown that these are associated with proarrhythmic changes on 12-lead electrocardiogram (ECG) and a higher risk of sudden cardiac death (SCD). However, these studies lack the deep electrophysiological phenotyping required to explain their observations. Electrocardiographic imaging (ECGi) is a non-invasive alternative to 12-lead ECG, by which epicardial potentials, electrograms and activation sequences can be recorded to study adverse electrophysiological modelling in greater depth and on a more focussed, subject-specific scale. Therefore, this study proposes to better define the risk of arrhythmia and understand the underlying adverse electrophysiological remodelling conferring this risk in three groups (obesity, RA and DCM). Firstly, data from two large, national repositories will be analysed to identify associations between routine clinical biomarkers and proarrhythmic 12-lead ECG parameters, to confirm adverse electrophysiological remodelling and a higher risk of arrhythmia. Secondly,ECGi will be performed before and after planned clinical intervention in obese and RA patients, and at baseline in titin-truncating variant (TTNtv)-positive and -negative DCM patients, to characterise the specific and potentially reversible conduction and repolarisation abnormalities that may underlie increased arrhythmic risk.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) occurs in groups that are neither traditionally considered high-risk nor have been the subject of large-scale studies. These include obesity, inflammatory arthropathy and gene-specific cardiomyopathy. Existing data to explain higher risk of arrhythmia in these cohorts rely on 12-lead ECG and therefore lack in-depth electrophysiological phenotyping. The investigators have access to the two large national data repositories providing a wealth of data to study risks of arrhythmia on a scale larger than any previously published study. They also have a proven track record of utilising electrocardiographic imaging (ECGi) to conduct in-depth investigation of electrophysiological remodelling to better characterise arrhythmic risk.

ECGi is a validated, noninvasive method of acquiring body surface potential data using 252-electrodes and combining it with subjectspecific heart-torso geometry from crosssectional imaging. Using inverse solution mathematical algorithms, the ECGi system reconstructs epicardial unipolar electrograms and panoramic activation and potential maps over a single sinus beat, which is visualised on a digitised image of the subject's heart. Various studies have demonstrated the efficacy of ECGi to localise ventricular arrhythmias; more accurately calculate QT interval dispersion than 12-lead ECGs in obesity; and characterise ventricular tachycardia (VT) with intramural re-entry following myocardial infarction-induced scarring.

The study aims to confirm that obesity, RA and DCM are risk factors for arrhythmia and associated with electrophysiological remodelling manifest on 12-lead ECG, using large data repositories. The investigators will also perform electrocardiographic imaging (ECGi) to investigate and understand specific, and potentially reversible, conduction and repolarisation abnormalities conferring risk of arrhythmia in these cohorts using ECGi.

Hypotheses:

1. Routine clinical biomarkers correlate with proarrhythmic 12-lead ECG parameters
2. Adverse (proarrhythmic) electrophysiological remodelling can be quantified with ECGi
3. Bariatric surgery reverses adverse electrophysiological remodelling in obesity
4. Pharmacological therapy reverses adverse electrophysiological remodelling in RA
5. TTNtv is associated with adverse electrophysiological remodelling in DCM

In-keeping with hypothesis 1, the study population will include participants from the UK biobank and Airwave Health Monitoring Study in which risk of arrhythmia will be defined. Participants in both data repositories provided informed consent for their data to be used for research.

With respect to hypotheses 2-5, the study will involve 3 distinct ECGi sub-studies, each in a well-defined cohort to identify specific, and potentially reversible, conduction and repolarisation abnormalities, and comparing the disease to healthy controls. These are:

i. Obesity (BMI >40) ii. RA iii. TTNtv-positive and -negative DCM

ELIGIBILITY:
Inclusion Criteria:

* patients with obesity (BMI>40) who will undergo stapled bariatric surgery
* RA, prior to commencement of disease-modifying drugs
* TTNtv-positive or -negative DCM
* no known existing medical condition or health concerns i.e. healthy volunteers;
* aged 18 to 75 years, inclusive

Exclusion Criteria:

* aged under 18 or over 75 years;
* known HIV, hepatitis B & C or vCJD infection;
* unable to provide verbal or signed written informed consent;
* pregnancy or positive urinary pregnancy test;
* breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients awaiting stapled bariatric surgery, without a history of or concomitant ischaemic or structural heart disease, arrhythmia or receiving anti-arrhythmic medication, will be recruited prospectively from the bariatric surgery preoperative assessment clinics.
  Similarly, patients with RA will be recruited prospectively from rheumatology clinics, prior to initiation of biologic or diseased modifying anti-rheumatic drugs. TTNtv-positive and -negative DCM patients an existing data registry will be recalled for this study. Healthy volunteers: will be recruited from our affiliated institutions who have given prior consent to be contacted for research.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Activation-recovery intervals | 30 months approximately ie at the end of the study
  Electrocardiographic parameter
Conduction velocity | 30 months approximately ie at the end of the study
  Electrocardiographic parameter

CONTACTS AND LOCATIONS:
Overall Officials: Fu Siong Ng, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Imperial College London (Hammersmith campus), London
  - St Mary's Hospital, London

IPD SHARING:
Plan to Share IPD: No
Only anonymised data will be shared amongst the research team. This includes electrocardiographic, imaging, demographic, biochemical and other clinical data.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT03910725/Prot_SAP_001.pdf
  • Informed Consent Form (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT03910725/ICF_000.pdf